CLINICAL TRIAL: NCT02898532
Title: The Influence of Participating in Target Shooting Sport on Inattentive, Hyperactive and Impulsive Symptoms in Children - A Controlled Study of Best Practice.
Brief Title: Children With ADHD and ADHD-like Symptoms and Target Shooting Sport in Danish Shooting Associations.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Annegrete Maansson, PhD-student, University of Southern Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SDU-SUN-VEK20130134
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: ADHD
Keywords: Children, ADHD, target shooting sport
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Active Comparator): The intervention is organised in collaboration between the local school, the Danish Shooting Association, and the national DGI (The Danish Gymnastics and Sporting Organization). The intervention is available geographical nationwide. The children will practise target-shooting sport in local Shooting Association once a week during school hours for a period of 6 months. Selected schools are either special schools or municipal schools with special educational programmes for children diagnosed with either ADHD or severe difficulties of hyperactivity, inattention and impulsivity. Teachers accompany the children to the Shooting Association where the instructors meet them.
  Interventions: Behavioral: Educational programmes
- Control group (No Intervention): The same target group as children in the intervention group. In the control group children are not practicing target shooting sport, neither in school or free time.

INTERVENTIONS:
Behavioral: Educational programmes — Children with ADHD or ADHD-like symptoms practicing target shooting sport in Danish Shooting Associations, during schooltime, for 6 months.
  Arms: Intervention group

SUMMARY:
Practising target shooting sport requires focused attention and motoric steadiness. Parental reports suggest that children with attention-deficit/hyperactivity disorder (ADHD) benefit from participating in target shooting sport in Danish Shooting Associations.

Aim: This study aims at examining if and to which extent target shooting sport in children with attention difficulties reduces parent- and teacher-reported severity of inattentiveness, hyperactivity, and impulsivity, and improves the children's well-being and quality of life.

DETAILED DESCRIPTION:
Children with Attention Deficit Hyperactivity Disorder (ADHD) (DSM-5) are characterised by three core symptoms: inattention, hyperactivity and impulsivity. Approximately 2-3 % of Danish school children are diagnosed with ADHD (Madsen, Ersbøll, Olsen, Parner, & Obel, 2015), and the prevalence in Denmark is about 5 % (Dalsgaard, Nielsen, & Simonsen, 2013). Many children with ADHD experience difficulties in managing social relations, e.g. team sports, and are often excluded from leisure activities with other children. This can have an impact on their well-being and quality of life which to a high degree depend on whether they have friends and communities with peers (Riley et al., 2006). Almost 50 % of children with ADHD experience the core symptoms in adulthood, and many develop psychological and social problems (Dalsgaard, Mortensen, Frydenberg, & Thomsen, 2013) and are at risk of premature death (Dalsgaard, Ostergaard, Leckman, Mortensen, & Pedersen, 2015). The NICE guideline (National Collaborating Centre for Mental Health, 2009) recommends a combination of pharmacological and psychosocial treatment (multimodal treatment approach) for children aged 6-18 years, to remedy other symptoms than ADHD core symptoms. A growing focus on the benefits of sports activities, yoga and mindfulness suggests that physical activity may have a positive impact on children and young people with ADHD (Cerrillo-Urbina et al., 2015; Kang, Choi, Kang, & Han, 2011; Haydicky, Wiener, Badali, Milligan , & Ducharme, 2012; van der Oord, Bogels, & Peijnenburg, 2012; van de Weijer-Bergsma, Formsma, de Bruin, & Bogels, 2012).

The sport of Target shooting can be regarded as a type of mental training in which the athlete uses techniques breathing to calm down, focus and improve attention. Mind and body must be in complete balance and the techniques used are similar to those used in meditation (Jeppesen & Pensgaard, 2006). Furthermore, regulations apply to the Danish Shooting Associations, in combination with the way the target shooting sport is practiced in Denmark is associated with fixed physical boundaries, clear rules and a distinct structure for the activity. Furthermore, it is a sport where the adult instructor always is very close to the child, and it is custom for the instructor gives instructions in a calm, structured and concise manner. Thus, target-shooting sport has implicitly features elements that can be considered protective environmental factors for the inattentive child and thus may contribute to reduce ADHD-symptoms and strengthen the child's well-being and quality of life. In 2012, the Danish Gymnastics and Sporting Organization (DGI) initiated a sports project, where children with ADHD or similar symptoms of inattention, hyperactivity and impulsivity practiced target-shooting sport in Danish Shooting Association. The evaluation showed, that the children became more concentrated and focussed during the training (Maansson, 2015). Based on this experience, this study has been initiated. However no studies have investigated the effect of target shooting sports for children with difficulties with inattention, hyperactivity and impulsivity.

The main aim of this study is therefore to investigate the influence of participation in target shooting sports in Danish Shooting Association for children having difficulties with inattention, hyperactivity and impulsivity.

ELIGIBILITY:
Inclusion Criteria:

Children following criteria: Age 10-14 years, either ADHD diagnosis or selected by school staff or school psychologist to show distinct difficulties with inattention, hyperactivity and impulsivity, which affects the child's school attendance. If the child receives pharmacological treatment for ADHD and the treatment is expected to be stable during the intervention period.

Exclusion Criteria:

Children showing a physical visual handicap or severe symptoms of current mental health difficulties such as psychosis or suicidal ideations or impulses are not included.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Teacher-rated ADHD-RS-IV. | Pre- and post (6 months after commencement) intervention
  The total score on the relevant 18 items on symptoms of inattention, hyperactivity and impulsivity on the teacher-rated ADHD-RS-IV.

SECONDARY OUTCOMES:
Qb-test. | Pre- and post (6 months after commencement) intervention
  Hyperactivity (distance and area) and inattention (reaction time variance and omission errors) as measured by the Qb-test.
Parent-rated ADHD-RS-IV. | Pre- and post (6 months after commencement) intervention
  The total score on the relevant 18 items on symptoms of inattention, hyperactivity and impulsivity on the parent-rated ADHD-RS-IV.
Teacher- and parent-rated SDQ. | Pre- and post (6 months after commencement) intervention
  The total scores on the teacher- and parent-rated SDQ.
Child-rated Kidscreen-27 | Pre- and post (6 months after commencement) intervention
  Quality of life as measured by the total score on the child-rated Kidscreen-27.
Interviews | Prior to intervention (1 month) start, during intervention period (6 months) and after end of intervention (1-3 months). A total period of 8-10 months.
  Semistructured qualitative Interviews with parents, teachers and children. Focus on children's participation and engagement and mechanisms of change.
Observations | Prior to intervention (1 month) start, during intervention period (6 months) and after end of intervention (1-3 months). A total period of 8-10 months.
  Observations of children (interventions group) in classroom and in the Shooting Association. Focus on participation and engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Kaya Roessler, Ph.D., Prof., Study Director — Department of Psychology.; Annegrete Maansson, Ph.D fellow, Principal Investigator — Department of Psychology.
Locations (1):
- Odense kommune, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mansson AG, Elmose M, Dalsgaard S, Roessler KK. The influence of participation in target-shooting sport for children with inattentive, hyperactive and impulsive symptoms - A controlled study of best practice. BMC Psychiatry. 2017 Mar 28;17(1):115. doi: 10.1186/s12888-017-1283-5. PMID 28351351